CLINICAL TRIAL: NCT07261280
Title: Testing a Biometric Identification System to Improve Malaria Vaccine Completion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Ghana (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Elisa Maria Maffioli, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00270320
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Vaccination
Keywords: Vaccine; Malaria; Adherence; Biometrics; Health Systems
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Health facilities randomized in treatment clusters will be provided with a digital vaccination record system (e-tracker) linked to biometrics (facial recognition) of caregivers (if child is below 6 months) or of children (if child is above 6 months) [HEALTH FACILITY INTERVENTION]. Caregivers (if child is below 6 months) or children (if child is above 6 months) living in communities in the catchment areas of health facilities randomized in treatment clusters [INDIVIDUAL INTERVENTION] will be registered at the community level into the e-tracker and biometrics (facial recognition), and caregivers of children who are due for or missed vaccination will receive voice message appointment reminders if they provided a phone number during the registration in biometrics.
  Interventions: Behavioral: HEALTH FACILITY INTERVENTION; Behavioral: INDIVIDUAL INTERVENTION
- Control (No Intervention): Health facilities randomized in control clusters, and caregivers (if child is below 6 months) or children (if child is above 6 months) living in communities in the catchment areas of health facilities randomized in control clusters will not receive any intervention during the study period.

INTERVENTIONS:
Behavioral: HEALTH FACILITY INTERVENTION — Health facilities randomized in treatment clusters will be provided with a digital vaccination record system (e-tracker) linked to biometrics (facial recognition) of caregivers (if child is below 6 months) or of children (if child is above 6 months). With the support of Ghana Health Services, Simprints will train CHWs on digital vaccination record system (e-tracker) and biometrics. Simprints will also provide Technical Assistance to CHWs for the duration of the study.
  Arms: Treatment
Behavioral: INDIVIDUAL INTERVENTION — Caregivers (if child is below 6 months) or children (if child is above 6 months) living in communities in the catchment areas of health facilities randomized in treatment clusters will be registered at the community level into the e-tracker and biometrics (facial recognition), and caregivers of children who are due for or missed vaccination will receive voice message appointment reminders if they provided a phone number during the registration in biometrics. Reminders will be sent before a child is due a visit to receive vaccination, as well as after a child missed his due visit.
  Arms: Treatment

SUMMARY:
Receiving all four doses of the malaria vaccine can significantly protect children against malaria illness, hospitalization, and death. However, in Ghana, only 46% of children complete the full vaccination sequence. More broadly, many children in Ghana do not receive the full set of recommended pediatric vaccinations. To address this, Simprints, in collaboration with Ghana Health Services, will implement a digital vaccination record system linked to biometrics. This system will automatically identify children who are behind on their vaccination schedule, providing health workers with information to prioritize community outreach. Additionally, it will send voice message reminders to caregivers to improve compliance. A cluster-randomized controlled trial (c-RCT) will be conducted in the Oti region to measure the impact of this innovation on the proportion of children completing malaria and routine vaccination schedules.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (in the last two trimesters), aged 15-49 years old, who do not plan to permanently move in the next 12 months.
* Women with children under 6 months old, aged 15-49 years old, who do not plan to permanently move in the next 12 months.

Exclusion Criteria:

* Non-age-eligible women.
* Men and non-emancipated minors.
* Women who do not consent.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female
Enrollment: 4715 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Completion of full malaria sequence (Index children) | Measured at endline, 24-26 months after baseline
  Record of 4 doses of malaria vaccines for the index child recorded by the individual child's booklet (or self-reported by the mother if the booklet is not available)
Timely full malaria vaccination (Index children) | Measured at endline, 24-26 months after baseline
  Record of 4 doses of malaria vaccines for the index child recorded by the individual child's booklet (or self-reported by the mother if the booklet is not available) taken within the appropriate time frame.
Completion of full routine vaccination sequence (basic antigens) (Index children) | Measured at endline, 24-26 months after baseline
  Records of doses of routine vaccines (basic antigens) for the index child recorded in the individual child's booklet (or self-reported by the mother if the booklet is not available). Defined as receipt of all of the following:
  One dose of BCG vaccine; Three doses of polio vaccine given as oral polio vaccine (OPV); Inactivated polio vaccine (IPV); Three doses of Pentavalent vaccine (Penta); One dose of measles-rubella vaccine (MR).
Completion of full routine vaccination sequence (national schedule) (Index children) | Measured at endline, 24-26 months after baseline
  Records of doses of routine vaccines (national schedule) for the index child recorded in the individual child's booklet (or self-reported by the mother if the booklet is not available).
  Full vaccination coverage based on the national schedule is defined as the index child having received all the following:
  BCG; Three doses of Pentavalent (Penta); Four doses of OPV (including OPV given at birth); One dose of IPV; One dose of yellow fever vaccine; Three doses of pneumococcal vaccine (PCV); Three doses of rotavirus vaccine; Two doses of measles-rubella vaccine (MR); One dose of meningitis A vaccine (MenA).

SECONDARY OUTCOMES:
Timely full routine vaccination sequence (basic antigens) (Index children) | Measured at endline, 24-26 months after baseline
  Records of doses of routine vaccines (basic antigens) for the index child recorded in the individual child's booklet (or self-reported by the mother if the booklet is not available). Taken within the appropriate time frame.
Timely full routine vaccination sequence (national schedule) (Index children) | Measured at endline, 24-26 months after baseline
  Records of doses of routine vaccines (national schedule) for the index child recorded in the individual child's booklet (or self-reported by the mother if the booklet is not available).
  Full vaccination coverage based on the national schedule is defined as the index child having received all the following, taken within the appropriate time frame.
Early, Late or Very Late malaria vaccination (Index children) | Measured at endline, 24-26 months after baseline
  Record of 4 doses of malaria vaccines for the index child recorded by the individual child's booklet (or self-reported by the mother if the booklet is not available). Taken outside the appropriate time frame.
Early, Late or Very Late full routine vaccination sequence (basic antigens) (Index children) | Measured at endline, 24-26 months after baseline
  Records of doses of routine vaccines (basic antigens) for the index child recorded in the individual child's booklet (or self-reported by the mother if the booklet is not available). Taken outside the appropriate time frame
Early, Late or Very Late full routine vaccination sequence (national schedule) (Index children) | Measured at endline, 24-26 months after baseline
  Records of doses of routine vaccines (national schedule) for the index child recorded in the individual child's booklet (or self-reported by the mother if the booklet is not available). Taken outside the appropriate time frame.
Number of malaria vaccines taken (Index children) | Measured at endline, 24-26 months after baseline
  Number of recorded malaria vaccines taken (from 0 to 4) by the index child recorded by the individual child's booklet (or self-reported by the mother if the booklet is not available).
Number of routine vaccines taken (basic antigens) (Index children) | Measured at endline, 24-26 months after baseline
  Number of recorded basic antigens taken (0 to 9) by the index child recorded by the individual child's booklet (or self-reported by the mother if the booklet is not available).
Number of routine vaccines taken (full national schedule) (Index children) | Measured at endline, 24-26 months after baseline
  Number of recorded vaccinations taken (0 to 19) from the national schedule by the index child recorded by the individual child's booklet (or self-reported by the mother if the booklet is not available)
Number of timely malaria vaccines taken (Index children) | Measured at endline, 24-26 months after baseline
  Number of recorded malaria vaccines taken (from 0 to 4) within the appropriate time frame by the index child recorded by the individual child's booklet (or self-reported by the mother if the booklet is not available).
Number of timely routine vaccines taken (basic antigens) (Index children) | Measured at endline, 24-26 months after baseline
  Number of recorded basic antigens taken (0 to 9) within the appropriate time frame by the index child recorded by the individual child's booklet (or self-reported by the mother if the booklet is not available)
Number of timely routine vaccines taken (full national schedule) (Index children) | Measured at endline, 24-26 months after baseline
  Number of recorded vaccinations taken (0 to 19) from the national schedule within the appropriate time frame by the index child recorded by the individual child's booklet (or self-reported by the mother if the booklet is not available)
Received each vaccine on time (full national schedule) (Index child), analyzed individually | Measured at endline, 24-26 months after baseline
  Among each of the following, analyzed individually, index child received the vaccine within the appropriate time frame according to the national schedule (as recorded in the individual child's booklet or as self-reported by the mother)
Up to date on malaria vaccine (children under 3 years old in study households) | Measured at endline, 24-26 months after baseline
  Record of having taken all doses of malaria vaccine as appropriate for child's age as recorded by the children's booklets (or self-reported by the mother if the booklet is not available)
Up to date on routine vaccines (basic antigens) (Children under 3 years old in study households) | Measured at endline, 24-26 months after baseline
  Record of having taken all doses of basic antigens as appropriate for child's age as recorded by the children' s booklets (or self-reported by the mother if the booklet is not available)
Up to date on routine vaccines (full schedule) (Children under 3 years old in study households) | Measured at endline, 24-26 months after baseline
  Record of having taken all doses of national vaccine schedule as appropriate for child's age as recorded by the children' s booklets (or self-reported by the mother if the booklet is not available)
Cumulative number of late days in receipt of malaria vaccination (index children) | Measured at endline, 24-26 months after baseline
  Among those who received at least a dose of the malaria vaccine, the number of days late the vaccine(s) were relative to what the national schedule considers "on time" for each dose. Late days are equal to zero for those who received the vaccine on time or early.
Cumulative number of late days in receipt of basic antigens (index children) | Measured at endline, 24-26 months after baseline
  Among those who received at least one dose of basic antigens, the number of days late the vaccine(s) were relative to what the national schedule considers "on time" for each dose. Late days are equal to zero for those who received the vaccine on time or early.
Cumulative number of late days in receipt of routine vaccines according to national schedule (index children) | Measured at endline, 24-26 months after baseline
  Among those who received at least one dose of routine vaccines according to the national schedule, the number of days late the vaccine(s) were relative to what the national schedule considers "on time" for each dose. Late days are equal to zero for those who received the vaccine on time or early.
Mother knows when to bring the child to the clinic for the first vaccination | Measured at endline, 24-26 months after baseline
  Mother self-reports being sure or very sure about when to bring the child to the clinic for the first vaccination
Facility Vaccine Data Accuracy | Measured around endline, 24-26 months after baseline
  Discrepancy in the total number of children vaccinated based on paper-based records at the facility vs digital records in DHMIS 2. Measured as the vaccine "verification factor" for BCG, Penta 3 and MR-2 over a three month period, comparing the total number of children vaccinated with each of the three vaccines over this period reported in DHIMS 2 with the paper-based record.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Maria Maffioli, PhD, Principal Investigator — University of Michigan; Jessica Cohen, PhD, Principal Investigator — Harvard University; Chris Guure, Principal Investigator — University of Ghana
Locations (1):
- Communities in Oti Region, Oti Region, Ghana

IPD SHARING:
Plan to Share IPD: No